CLINICAL TRIAL: NCT05220488
Title: Fear of COVID-19 and Physical Activity Level of Children With Asthma
Brief Title: Fear of COVID-19 and Physical Activity in Children With Asthma During the Covid Period
Status: Completed | Type: Observational
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Şeyma Nur Önal, Lecturer, Bartın Unıversity
Other Study IDs: COVID-19asthmachildphysicalact
Record Dates: First submitted 2022-01-29; First posted 2022-02-02 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Asthma in Children
Keywords: Asthma; COVID-19; Physical Activity
MeSH Terms: conditions — Asthma; COVID-19; Motor Activity | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma Group: Asthma Group
  Interventions: Other: Assessment
- Healthy Group: Healthy Group
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Parameters such as physical activity and fear of covid will be evaluated in asthmatic and healthy children and adolescents.

SUMMARY:
Social isolation rules applied to prevent and control COVID-19 disease reduce cross-infection, exposure to more allergens in the home environment, reducing hospital admissions by avoiding contamination, asthma control, fear of COVID-19 and physical activity for reasons such as increased anxiety and lack of exercise. How it will affect is unclear. Considering all these, positive or negative changes in asthma-related risk factors, changes in physical activity level, asthma attacks and control, fear of COVID-19 will be examined and contribute to the literature in children with asthma.

DETAILED DESCRIPTION:
Social isolation rules applied to prevent and control COVID-19 disease reduce cross-infection, exposure to more allergens in the home environment, reducing hospital admissions by avoiding contamination, asthma control, fear of COVID-19 and physical activity for reasons such as increased anxiety and lack of exercise. How it will affect is unclear. Considering all these, positive or negative changes in asthma-related risk factors, changes in physical activity level, asthma attacks and control, fear of COVID-19 will be examined and contribute to the literature in children with asthma. Therefore, our primary aim in our study is; The aim of this study is to examine the asthma control and COVID-19 fear levels of asthmatic children who were in social isolation during the COVID-19 pandemic in children with asthma and compare their effects compared to healthy children. Our secondary aim in our study; The aim of this study is to examine the physical activity levels of children in social isolation during the COVID-19 pandemic in children with asthma.

Asthma Group Inclusion Criteria:

* Having been diagnosed with asthma,
* In addition, not having any chronic disease,
* Volunteering to participate in the study,
* Not having speech and hearing problems,
* Being cooperative,
* Not having mental, neurological, orthopedic, cardiovascular or pulmonary problems that would prevent physical activity,

Asthma Group Exclusion Criteria:

* The presence of a medical indication that requires complete restriction of physical activity,
* To have had COVID-19 in the last 1 month or to be newly diagnosed with COVID-19,
* Having symptoms of COVID-19 and suspected illness,
* Existence of cooperation and communication problems.

Healthy Group Inclusion Criteria

* Not having any chronic disease for healthy individuals,
* Volunteering to participate in the study,
* Not having speech and hearing problems,
* Being cooperative,
* Not having a mental, neurological, orthopedic, cardiovascular or pulmonary problem that would prevent physical activity,

Healthy Group Exclusion Criteria

* The presence of a medical indication that requires complete restriction of physical activity,
* To have had COVID-19 in the last 1 month or to be newly diagnosed with COVID-19,
* Having symptoms of COVID-19 and suspected illness,
* Existence of cooperation and communication problems

ELIGIBILITY:
Inclusion Criteria:

* Asthma Group Inclusion Criteria:
* Having been diagnosed with asthma,
* In addition, not having any chronic disease,
* Volunteering to participate in the study,
* Not having speech and hearing problems,
* Being cooperative,
* Not having mental, neurological, orthopedic, cardiovascular or pulmonary problems that would prevent physical activity,

Healthy Group Inclusion Criteria

* Not having any chronic disease for healthy individuals,
* Volunteering to participate in the study,
* Not having speech and hearing problems,
* Being cooperative,
* Not having a mental, neurological, orthopedic, cardiovascular or pulmonary problem that would prevent physical activity,

Exclusion Criteria:

* Asthma Group Exclusion Criteria:
* The presence of a medical indication that requires complete restriction of physical activity,
* To have had COVID-19 in the last 1 month or to be newly diagnosed with COVID-19,
* Having symptoms of COVID-19 and suspected illness,
* Existence of cooperation and communication problems. Healthy Group Inclusion Criteria
* Not having any chronic disease for healthy individuals,
* Volunteering to participate in the study,
* Not having speech and hearing problems,
* Being cooperative,
* Not having a mental, neurological, orthopedic, cardiovascular or pulmonary problem that would prevent physical activity,

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Asthmatic and healthy children and adolescents
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Physical Activity Questionnaire | 10 minutes
  It will be evaluated by Physical Activity Questionnaire-Child and Physical Activity Questionnaire-Adolescent. The scale consists of 10 questions and item 10 questions the presence of an illness or an acute condition that limits physical activity. Frequent activities (hopping, walking, football, gymnastics, dance, etc.), level of participation in physical education class, and frequency of activities during break time, lunch time, after school, evening hours and weekends, during leisure time in the last seven days The frequency of the activities performed and the frequency of sports, dance, games and other similar physical activities seven days a week are questioned.

SECONDARY OUTCOMES:
Asthma Control Test | 5 minutes
  Asthma Control Test: The Asthma Control Test (AKT) was developed to evaluate people's asthma control. It consists of 5 questions. It is applied to children over 12 years old. Questions are scored between 1-5. A minimum of 5 points and a maximum of 25 points are taken. If the total score is 25, it is considered as complete control, 24-20 as partial control, and ≤19 as not under control (17). In the 2020 Asthma Guide update, the total score is defined as 5-15 uncontrolled asthma, 16-19 insufficient control, 20-25 good control. Uysal et al. The Cronbach's alpha value of the scale, whose validity and reliability in Turkish was made by Dr., was found to be 0.84 (18). It will be used in the form to be applied to adolescents.
Fear of COVID-19 | 5 minutes
  Qualitative Questions on Examining the Fear of COVID-19:
  1. I am very afraid of the coronavirus (Covid-19).
  2. I am afraid of dying from coronavirus.
  3. I can't sleep because of the fear of catching the coronavirus.
  10. I am afraid of catching coronavirus and being hospitalized.
Social Isolation | 4 weeks
  Social Isolation
  1. In the last 4 weeks, how many days have participants been out of the house outdoors? (park, nature, field, garden, etc.)
  2. In the last 4 weeks, how many days have participants been out of the house indoors? (shopping mall, workplace, market, home visit etc.)
  3. In the last 4 weeks, how many days has an outsider come to participants r home? (Guest, relative, etc.)
  4. In the last 4 weeks, how many days has someone from the house outside of participants went out of the house? (park, nature, field, garden, etc.)
  5. In the last 4 weeks, how many days has someone other than participants gone out of the house indoors? (shopping mall, workplace, market, home visit etc.)
  6. In the last 4 weeks, I have warned family members who have come from outside to wash their hands and faces before removing their masks.
  Questions; Never, 1-3 days, 4-7 days, 7-15 days, 16-22 days, 23-30 days will be answered. The questions were created by the researchers.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma Nur Önal, Principal Investigator — Bartın Unıversity
Locations (1):
- Bartın University, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rothan HA, Byrareddy SN. The epidemiology and pathogenesis of coronavirus disease (COVID-19) outbreak. J Autoimmun. 2020 May;109:102433. doi: 10.1016/j.jaut.2020.102433. Epub 2020 Feb 26. PMID 32113704
- [Result] Skevaki C, Karsonova A, Karaulov A, Xie M, Renz H. Asthma-associated risk for COVID-19 development. J Allergy Clin Immunol. 2020 Dec;146(6):1295-1301. doi: 10.1016/j.jaci.2020.09.017. Epub 2020 Sep 28. PMID 33002516
- [Result] Lovinsky-Desir S, Deshpande DR, De A, Murray L, Stingone JA, Chan A, Patel N, Rai N, DiMango E, Milner J, Kattan M. Asthma among hospitalized patients with COVID-19 and related outcomes. J Allergy Clin Immunol. 2020 Nov;146(5):1027-1034.e4. doi: 10.1016/j.jaci.2020.07.026. Epub 2020 Aug 6. PMID 32771560
- [Result] Barsoum Z. Pediatric Asthma & Coronavirus (COVID-19)-Clinical Presentation in an Asthmatic Child-Case Report. SN Compr Clin Med. 2020;2(6):700-702. doi: 10.1007/s42399-020-00310-3. Epub 2020 May 19. PMID 32838131
- [Result] Papadopoulos NG, Custovic A, Deschildre A, Mathioudakis AG, Phipatanakul W, Wong G, Xepapadaki P, Agache I, Bacharier L, Bonini M, Castro-Rodriguez JA, Chen Z, Craig T, Ducharme FM, El-Sayed ZA, Feleszko W, Fiocchi A, Garcia-Marcos L, Gern JE, Goh A, Gomez RM, Hamelmann EH, Hedlin G, Hossny EM, Jartti T, Kalayci O, Kaplan A, Konradsen J, Kuna P, Lau S, Le Souef P, Lemanske RF, Makela MJ, Morais-Almeida M, Murray C, Nagaraju K, Namazova-Baranova L, Garcia AN, Yusuf OM, Pitrez PMC, Pohunek P, Pozo Beltran CF, Roberts GC, Valiulis A, Zar HJ; Pediatric Asthma in Real Life Collaborators. Impact of COVID-19 on Pediatric Asthma: Practice Adjustments and Disease Burden. J Allergy Clin Immunol Pract. 2020 Sep;8(8):2592-2599.e3. doi: 10.1016/j.jaip.2020.06.001. Epub 2020 Jun 17. PMID 32561497